CLINICAL TRIAL: NCT06718504
Title: The Effect of Virtual Reality Glasses on Pain, Anxiety, and Comfort During Upper Gastrointestinal System Endoscopy: Randomized Controlled Trial
Brief Title: The Effect of Virtual Reality Glasses During Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Elif Gezginci, Assoc. Prof., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 167
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Pain; Anxiety; Gastro-Intestinal Disorder
Keywords: Pain; Anxiety; Comfort; Endoscopy; Virtual Reality Glasses
MeSH Terms: conditions — Pain; Anxiety Disorders; Digestive System Diseases

STUDY DESIGN:
Intervention Model Description: This study is a single-center parallel-group randomized controlled clinical trial. Participants who met the inclusion criteria for the study were divided into two equal groups: the intervention group (n=30) and the control group (n=30).
  according to the computer-based randomization table.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): During the procedure, patients in the intervention group watched videos of their choice, either in a relaxing natural setting or without any violent content, using virtual reality glasses.
  Interventions: Device: Virtual Reality Glasses
- Control Group (No Intervention): No intervention was applied to the patients in the control group.

INTERVENTIONS:
Device: Virtual Reality Glasses — Virtual reality is a method that can be used to distract and prepare patients for medical procedures. Virtual reality is a computer-generated environment where three-dimensional interaction is possible. It is an advanced technology that allows an individual to move into a virtual environment and focus their attention on other thoughts, allowing them to pay less attention to pain and anxiety. In this study, the virtual reality glasses were put on for the intervention group five minutes before the procedure began and were kept on until the procedure was completed. The virtual reality glasses showed the patient-selected images of a relaxing nature setting or images without any violent content.
  Arms: Intervention Group

SUMMARY:
Upper gastrointestinal endoscopy is an invasive procedure used to diagnose and treat pathologies in the gastrointestinal mucosa. Since it is an invasive procedure, it can cause anxiety in patients before and pain during the procedure. Virtual reality glasses are an effective method used to reduce the pain and anxiety levels of patients during painful procedures. This study aimed to evaluate the effects of virtual reality glasses on pain, anxiety, and comfort in patients undergoing upper gastrointestinal endoscopy without sedation.

DETAILED DESCRIPTION:
This single-center randomized controlled parallel group study was conducted with 60 patients who underwent upper gastrointestinal endoscopy at the Endoscopy Unit of a training and research hospital in Istanbul. Patients in the virtual reality glasses group (n=30) watched videos of their preferred relaxing nature settings or videos without any violent content during the procedure. Patients in the control group (n=30) received no intervention. Data were collected using the Patient Information Form, Visual Analog Scale (for pain and comfort) and State Anxiety Inventory. Pain, comfort and anxiety levels of patients were assessed five minutes before and five minutes after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* To have an upper gastrointestinal endoscopy for the first time
* To be performed an upper GI endoscopy without sedation
* To be between the ages of 18-75
* To be willing to participate in research

Exclusion Criteria:

* To use analgesic or anesthetic drugs before or during the procedure
* To use antidepressants, anxiolytic and sedative drugs
* To have communication difficulties and mental disability

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Change on pain intensity as measured by Visual Analog Scale | five minutes before endoscopy and five minutes after endoscopy
  The average score change on pain intensity as measured by Visual Analog Scale. This scale is an unidimensional measure commonly used to measure pain intensity. The scale is a measuring tool with length of 0-10 cm. High scores on the scale indicate that pain intensity is high.

SECONDARY OUTCOMES:
Change on anxiety level as measured by State-Trait Anxiety Inventory | five minutes before endoscopy and five minutes after endoscopy
  The average score change on anxiety level as measured by State-Trait Anxiety Inventory. This scale in used to measure anxiety. The scores on the scale ranges from 20 to 80. The high scores on the scale indicate that anxiety is high.

OTHER OUTCOMES:
Change on satisfaction level as measured by Visual Analog Scale | five minutes before endoscopy and five minutes after endoscopy
  The average score change on satisfaction level as measured by Visual Analog Scale. This scale is an unidimensional measure commonly used to measure satisfaction level. The scale is a measuring tool with length of 0-10 cm. High scores on the scale indicate that satisfaction level is high.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Gezginci Akpınar, Assoc Prof, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Saglik Bilimleri Universitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No